CLINICAL TRIAL: NCT03100773
Title: Impact of Atraumatic Restorative Treatment Associated With Oral Health Educational Strategy on Dental Anxiety, Oral Health-related Quality of Life and Salivary Biochemical and Microbiological Characteristics of Brazilian Schoolchildren
Brief Title: Impact of Atraumatic Restorative Treatment and Oral Health Promotion on Psychological and Salivary Aspects of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Taís de Souza Barbosa, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJK-2014-ART
Record Dates: First submitted 2016-01-22; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Dental Caries
Keywords: alpha-amylases; child; cortisol; dental anxiety; dental atraumatic restorative treatment; health education; microbiota; oral hygiene; quality of life; saliva
MeSH Terms: conditions — Dental Caries; Health Education | interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group control (Experimental): Caries-free children submitted to four consecutive sessions of oral health educational strategy (once a week).
  Interventions: Other: Oral health educational strategy
- Group of strategy + ART (Experimental): Children with at least one decayed primary molar in dentin submitted to four consecutive sessions of oral health educational strategy (once a week) followed by Atraumatic Restorative Treatment (ART)
  Interventions: Other: Oral health educational strategy; Procedure: Atraumatic Restorative Treatment
- Group of ART (Experimental): Children with at least one decayed primary molar in dentin submitted to Atraumatic Restorative Treatment (ART)
  Interventions: Procedure: Atraumatic Restorative Treatment

INTERVENTIONS:
Other: Oral health educational strategy — Oral health educational strategy consisted of four consecutive sessions (once a week) about etiological factors of caries (using visual aids), oral hygiene instructions (using models), supervised toothbrushing and explanation of atraumatic restorative treatment (indications and stages).
  Arms: Group control; Group of strategy + ART
Procedure: Atraumatic Restorative Treatment — Atraumatic Restorative Treatment was performed using hand instruments for opening and cleaning the cavities and a high-viscosity glass-ionomer for restoration.
  Arms: Group of ART; Group of strategy + ART

SUMMARY:
This study evaluated the impact of atraumatic restorative treatment associated with oral health educational strategy on dental anxiety, oral health-related quality of life and salivary biochemical and microbiological characteristics of Brazilian schoolchildren.

DETAILED DESCRIPTION:
Children aged six- to eight years-old, both gender, were selected from public schools of Piracicaba, SP, Brazil, and were divided in three groups: caries-free children (control group, GC), children with at least one primary molar with dentin caries lesion submitted to oral health educational strategy followed by ART (GS+ART), and the other group was directly submitted to ART (GART). Oral hygiene was assessed by the presence of biofilm and gingivitis in buccal surfaces of primary and/or permanent upper incisors. Oral health educational strategy consisted of four consecutive sessions (once a week) about etiological factors of caries (using visual aids), oral hygiene instructions (using models), supervised toothbrushing and explanation of ART (indications and stages). ART was performed using hand instruments for opening and cleaning the cavities and a high-viscosity glass-ionomer for restoration. Dental anxiety was assessed by measuring the cognitive (modified Venham Picture Test, m-VPT), behavioral (modified Venham Anxiety Scale, m-VAS) and physiological (heart rate, HR; salivary cortisol and alpha-amylase, SC and SAA) aspects in the following days and moments: D1 - baseline, a day preceding ART (SC and SAA); D2 - day of treatment, before strategy (m-VPT), before ART (m-VPT, HR, SC, SAA), during the explanation of procedure (HR, m-VAS), at the moment of deepest excavation (HR, m-VAS), at the moment the restoration was applied (HR, m-VAS), after ART (m-VPT, HR, SC, SAA). The following variables were evaluated in three moments: T1 - baseline, T2 - one week after strategy (for both GC and GART) and T3 - one month after the strategy or ART for GC and GART, respectively. Oral health-related quality of life was assessed using Brazilian short version of the Child Perceptions Questionnaire (16-CPQ8-10) with 16 items. Salivary flow rate was estimated by chewing 0.3g of an inert and tasteless material, for approximately 70 cycles/min and spitting all the saliva produced for five minutes into a cooled tube. Salivary pH was determined immediately after collection, using a portable pH-meter. Salivary buffer capacity was performed by adding 1.5 ml of HCl/5 mM to a tube containing 0.5 mL of stimulated saliva. For detection and quantification of S. mutans, the microbial DNA in unstimulated saliva samples was isolated and subjected to quantitative PCR reactions (qPCR).

ELIGIBILITY:
Inclusion Criteria:

* caries-free;
* presence of at least one primary molar with dentin caries lesion (without painful symptoms, mobility and abscess).

Exclusion Criteria:

* indication for tooth extraction;
* presence of fistula;
* abscess or spontaneous toothache;
* insufficient tooth structure to support restoration;
* current use of medications that could interfere with the central nervous system;
* inappropriate behavior and/or refusal to participate.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in dental anxiety assessed by measuring the cognitive and behavioral aspects. | T1: one day preceding the oral health educational strategies (GS+ART) (m-VPT); T2: during ART procedure (GS+ART and GART) (m-VAS) and immediately after ART (GS+ART and GART) (m-VPT); T3: 10 minutes after ART (GS+ART and GART) (m-VPT).
  The cognitive and behavioral aspects were assessed by modified Venham Picture Test (m-VPT) and modified Venham Anxiety Scale (m-VAS), respectively (scores).
Change in dental anxiety assessed by measuring the salivary biomarkers. | T1: 30 min preceding the ART (GART) and one day preceding OHES (GS+ART); T2: immediately after ART (GS+ART/GART); T3: 10 min after ART (GS+ART/GART).
  The hormonal biomarker was assessed by saliva collection for cortisol - sC (in microgram per using commercially available kit (Salimetrics, State College, PA, USA) according to the manufacturer's directions.
Change in dental anxiety assessed by measuring the salivary biomarkers. | T1: 30 min preceding the ART (GART) and one day preceding OHES (GS+ART); T2: immediately after ART (GS+ART/GART); T3: 10 min after ART (GS+ART/GART).
  The enzymatic biomarker was assessed by saliva collection for alpha-amylase - sAA (in international units per milliliter of saliva - U/ml) using commercially available kit (Salimetrics, State College, PA, USA) according to the manufacturer's directions.
Change in dental anxiety assessed by measuring the physiological aspect. | T1: 30 min preceding the ART (GART) and one day preceding OHES (GS+ART); T2: during ART procedure (GS+ART/GART) and immediately after ART (GS+ART/GART); T3: 10 min after ART (GS+ART/GART).
  The physiological aspect was assessed by heart rate (HR, in beats per minute, bpm) using a digital monitor (S625x, Polar, Finland).
Change in salivary physicochemical properties. | T1: 1 week before oral health strategy (GC and GS+ART); T2: 1 week after oral health strategy (GC and GS+ART); T3: 1 month after oral health strategy (GC) and 1 month after ART (GS+ART).
  The physicochemical properties of saliva were measured by flow rate (mL/min), pH and buffer capacity. Salivary stimulated and unstimulated flow rates were estimated as the volume of saliva secreted per min (mL/min). Salivary pH was determined immediately after collection in stimulated saliva, using a portable pH-meter (Orion 3 Star Benchtop, Thermo Electron Corporation, USA). Buffer capacity was performed by adding 1.5 ml of 5 mM HCl to a tube containing 0.5 mL of stimulated saliva and further determination of salivary pH.
Change in salivary microbiological properties. | T1: 1 week before oral health strategy (GC and GS+ART); T2: 1 week after oral health strategy (GC and GS+ART); T3: 1 month after oral health strategy (GC) and 1 month after ART (GS+ART).
  The microbiological characteristics of saliva were measured by total bacteria and S. mutans levels. The detection and quantification of S. mutans and total bacteria, the microbial DNA in unstimulated saliva samples was isolated and subjected to quantitative PCR reactions (qPCR).

SECONDARY OUTCOMES:
Change in oral hygiene. | T1 : 1 week before oral health strategy (GC and GS+ART) and 30 min before ART (GART); T2: 1 week after oral health strategy (GC and GS+ART); T3: 1 week after ART (GART and GS+ART); T4: 1 month after ART (GART and GS+ART).
  Oral hygiene was assessed by the presence of biofilm and gingivitis in buccal surfaces of primary and/or permanent upper incisors (presence/absence; frequencies) (in scores).
Change in oral health-related quality of life. | T1: 1 week before oral health strategy (GC and GS+ART) and 30 min before ART (GART); T2: 1 week after oral health strategy (GC and GS+ART); T3: 1 week after ART (GART and GS+ART); T4: 1 month after ART (GART and GS+ART).
  Oral health-related quality of life was assessed using the Brazilian short version of the Child Perceptions Questionnaire (16-CPQ8-10), with 16 items (in scores).

CONTACTS AND LOCATIONS:
Overall Officials: Taís S Barbosa, PhD, Principal Investigator — University of Campinas, Brazil

IPD SHARING:
Plan to Share IPD: Undecided